CLINICAL TRIAL: NCT00480974
Title: Long Term Follow up in Sickle Cell Patients Treated by Hydroxyurea.Observational Retrospective Study.
Brief Title: Long Term Follow up in Sickle Cell Patients Treated by Hydroxyurea
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Dr Koren Ariel, Pediatric Hematology Unit - HaEmek Medical Center - Afula - Israel
Other Study IDs: 5321006.EMC
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Sickle Cell Anemia; Sickle Cell Thalassemia
Keywords: Sickle cell anemia; Sickle cell thalassemia; Hydroxyurea
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with Sickle cell anemia treated by Hydroxyurea
  Interventions: Other: Clinical follow up and laboratory analysis

INTERVENTIONS:
Other: Clinical follow up and laboratory analysis — Clinical follow up and laboratory analysis

SUMMARY:
Hydroxyurea was found to be a good treatment in adult patients with sickle cell anemia with significant decrease in the frequency of vaso-occlusive crises and other crises related to SCA. Several studies were published with relative short term follow up in pediatric and young adult age. The purpose of this study is to assess the long term follow up in a group of patients that initiated Hydroxyurea treatment in childhood.

DETAILED DESCRIPTION:
Hydroxyurea was found to be a good treatment in adult patients with sickle cell anemia with significant decrease in the frequency of vaso-occlusive crises and other crises related to SCA. Several studies were published with relative short term follow up in pediatric and young adult age. The purpose of this study is to assess the long term follow up in a group of patients that initiated Hydroxyurea treatment in childhood.

A long term follow up will be recorded in a cohort of twenty SCA patients treated by Hydroxyurea for a period between 5 to 12 years. The frequency of vaso-occlusive crises, acute chest syndrome, blood transfusions, and hospitalization will be recorded retrospectively. Also the mean hgb level and hgb F percentage will be summarized.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated by Hydroxyurea in the Pediatric Hematology Unit.

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Sickle Cell Anemia treated at the Pediatric Hematology Unit and receiving Hydroxyurea
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Study Director — Pediatric Hematology Unit, Ha'Emek Medical Center; Carina Levin, MD, Study Chair — Pediatric Hematology Unit - Ha'Emek Medical Center; Miri Golan, Student, Principal Investigator — Pediatric Hematology Unit - HaEmek Medical Center; Luci Zalman, PhD, Study Chair — Hematology Laboratory - HaEmek Medical Center
Locations (1):
- Pediatric Hematology Unit - HaEmek Medical Center, Afula, Israel